CLINICAL TRIAL: NCT07133815
Title: A Multicenter, Single Arm, Open Label Phase II Clinical Study Evaluating the Long-term Efficacy and Safety of SHR-1918 in Homozygous Familial Hypercholesterolemia Patients
Brief Title: Evaluate the Long-term Efficacy and Safety of SHR-1918 in Patients With Homozygous Familial Hypercholesterolemia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Suncadia Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1918-205
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Homozygous Familial Hypercholesterolemia
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1918 (Experimental)
  Interventions: Drug: SHR-1918

INTERVENTIONS:
Drug: SHR-1918 — SHR-1918

SUMMARY:
A multicenter, single arm, open label phase II clinical study evaluating the long-term efficacy and safety of SHR-1918 in homozygous familial hypercholesterolemia patients

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Subjects who received and completed the SHR-1918-301 study treatment in previous studies and were deemed to have therapeutic benefits by the researchers

Exclusion Criteria:

1. Known to be allergic to the investigational drug or any component of the investigational drug, or to have experienced severe allergic reactions to other antibody drugs;
2. History of malignant tumors in the past 5 years;
3. There are serious concurrent diseases
4. Pregnant or lactating women;
5. The researchers determined that the subjects had poor compliance or any inappropriate factors for participating in this trial

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of adverse events | during the study period About 48 months，

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Second Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided